CLINICAL TRIAL: NCT04878601
Title: Innovative Strategies to Increase ART Initiation and Viral Suppression Among HIV-positive Men in Malawi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Partners in Hope, Inc. (Industry); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Kathryn L. Dovel, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K01TW011484 (NIH); K01TW011484 (NIH)
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Hiv
Keywords: HIV; HIV Self-Testing; HIVST; Index HIVST; Index Testing; Men; Male Partners; Antiretroviral therapy; ART initiation; Home-based ART; ART retention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hbART (Experimental): Home-Based ART initiation and continuation for 3-months with male-specific counseling and assisted facility navigation at 4-months.
  Interventions: Other: Home-Based ART
- fbART (Active Comparator): Facility-Based ART initiation and continuation with male-specific counseling.
  Interventions: Other: Facility-Based ART

INTERVENTIONS:
Other: Home-Based ART — Healthcare provider will ask ART client for permission to conduct a home visit with their HIV+ partner. Providers will conduct a home visit with HIV+ partners to provide confirmatory HIV testing and ART initiation with a 30-day supply. Monthly home-based ART follow-up visits with male-specific messaging and 30-day supply distribution will take place for 3-months. At 4-months providers will provide assisted linkage to a nearby facility to join the facility-based ART program. Additional counseling will be provided.
  Arms: hbART
Other: Facility-Based ART — Healthcare provider will ask ART client for permission to conduct a home visit with their HIV+ partner. Providers will conduct a home visit with HIV+ partners to provide confirmatory HIV testing and assisted linkage to a nearby facility for facility-based ART initiation and continuation. Male clients will receive a 30-day supply each visit and return monthly.
  Arms: fbART

SUMMARY:
Men in Sub-Saharan Africa are less likely to test for HIV, initiate ART, and more likely to initiate ART at later stages of disease. Two overarching barriers keep HIV-positive men from accessing ART services: 1) Lack of male-friendly services, and 2) harmful gender norms. Home-based ART may improve ART initiation and retention among male partners who test HIV-positive through Index HIV self-testing (HIVST). We will pilot an intervention that provides home-based ART initiation and home-based continuation for 3-months, followed by assisted linkage to facility-based care at 4-months. 470 participants will be enrolled [209 females, 261 males]

DETAILED DESCRIPTION:
Men in Sub-Saharan Africa are less likely to test for HIV, initiate ART, and more likely to initiate ART at later stages of disease. Achieving epidemic control requires immediate, concentrated effort to engage this largely unreached population. Index partner testing, whereby partners of HIV-positive clients are refereed for HIV testing, is critical to identifying undiagnosed men and has been adopted as a national policy by the Malawi Ministry of Health because of its high acceptability and its dramatic increase on HIV testing uptake. Two overarching barriers keep HIV-positive men from accessing ART services: 1) Lack of male-friendly services, and 2) harmful gender norms. Home-based ART may improve ART initiation and retention among male partners who test HIV-positive through Index HIVST. We will pilot an intervention that provides home-based ART initiation and home-based continuation for male partners identified as HIV-positive through Index HIVST for 3-months, followed by assisted linkage to facility-based care at 4-months. This intervention offers opt-out ART and in-depth, male-specific counseling for 3-months before linking men to facility based care. We will directly compare home-based ART to facility-based ART, whereby a health care worker will conduct a home-visit with HIV+ male partners to provide confirmatory HIV testing and immediate assisted linkage to a nearby facility for facility-based ART initiation and continuation.

ELIGIBILITY:
Female Partner Inclusion Criteria:

* Male partner ≥15 years of age
* No reported interpersonal violence (IPV) as defined by World Health Organization (WHO) with the above male partner in the past 12-months
* Male partner ever tested HIV-positive
* Male partner not currently engaged in ART services, defined as:

  * Tested HIV-positive ≥14 days and not on ART ≥14 days after testing HIV- positive;
  * ≥14 days late for the first four-week follow up appointment; or
  * Initiated ART but ≥60 days late for last ART appointment;
  * Male partner living inside the facility catchment area (defined as any area that Healthcare Workers (HCWs) from the study facility routinely visit for tracing purposes)

Female Partner Exclusion Criteria:

* Male partner <15 years of age
* Reported interpersonal violence (IPV) as defined by WHO with the above male partner in the past 12-months
* Male partner never tested HIV positive
* Male partner tested HIV-positive <14 days ago
* Male partner currently engaged in ART services, defined as:

  * Initiated ART <14 days late for the first four-week follow up appointment
  * Initiated ART and <60 days late for last ART appointment
  * Male partner living outside the facility catchment area (defined as any area that HCWs from the study facility routinely visit for tracing purposes)

Men Living with HIV Inclusion Criteria:

* ≥15 years of age
* Tested HIV positive using Ministry of Health standard algorithm (Determine + Unigold)
* Not currently engaged in ART services, defined as:

  * Tested HIV-positive ≥14 days and not on ART ≥14 days after testing HIV-positive;
  * ≥14 days late for the first four-week follow up appointment; or
  * Initiated ART but ≥60 days late for last ART appointment;
  * Has not taken ART in the past 7-days, as indicated by a point of care (POC) urine assay
  * Living inside the facility catchment area (defined as any area that HCWs from the study facility routinely visit for tracing purposes)

Men Living with HIV Exclusion Criteria:

* <15 years of age
* Never tested HIV positive using Ministry of Health standard algorithm (Determine + Unigold)
* Tested HIV-positive <14 days ago
* Currently engaged in ART services, defined as:

  * Initiated ART
  * <14 days late for the first four-week follow up appointment
  * Initiated ART and <60 days late for last ART appointment
  * Has taken ART in the past 7-days, as indicated by a point of care (POC) urine assay
  * Living outside the facility catchment area (defined as any area that HCWs from the study facility routinely visit for tracing purposes)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 470 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Men's ART Initiation | 6 months
  ART initiation within 6-months of enrollment. Sourced from medical chart reviews.

SECONDARY OUTCOMES:
Men's 6-month Retention | 6 months
  6-month retention (<60 days ever late for ART). Sourced from medical chart reviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Partners in Hope, Lilongwe, Malawi